CLINICAL TRIAL: NCT00173420
Title: Mechanisms of Neuropathic Pain: Investigation by Contact Heat Evoked Potential
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700654
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2007-10-23 (Estimated); Status verified 2005-06

CONDITIONS: Peripheral Nerve Diseases
Keywords: Normal Controls
MeSH Terms: conditions — Peripheral Nervous System Diseases

SUMMARY:
In order to clarify the normal components of thermal and painful evoked potentials by heat in normal subjects of both genders and different age group, to clarify the effect of specific anatomy in pain transduction, transmission and modification, and to establish the effect of peripheral nerve and their terminal free ending on the nociceptive transduction, the investigators will use heat stimulation on normal controls and patients with neurological diseases to clarify such issues.

DETAILED DESCRIPTION:
Only a few studies focus on clinical diseases like neuropathic pain or neurogenic pain. Little is known about the differences between normal and pathogenic pain processing. It is an opportunity to apply EEG, ERPs in the clinical fields. In many clinical conditions, brain lesions provide a chance to study the possible roles of one neural structure in pain integration and processing. In addition the applications of EEG/ERPs on clinical conditions may be help in the understanding about mechanism and genesis of pain in pathogenic conditions, the diagnosis of pathogenic pain, and the therapeutic aspects of these abnormal pain senses.

One limit in the study of human pain is the inappropriate stimulation method. Evoked potentials by contact heat have previously been difficult to elicit due to slow temperature rise times associated with thermal stimulators. However recently, the CHEPS (Contact Heat-Evoked Potential Stimulator) is developed, which uses a newly developed heat-foil technology and can create a rapid heating rate (up to 70°C/sec). The baseline and peak temperature and the rising time can be precisely controlled. It provides a non-invasive technique in the investigation of human pain activation related to thermal and nociceptive pathways involved in pain processing. Unlike the heat stimulation delivered by laser, CHEPS can deliver noxious thermal stimuli repeatedly to a large area of skin to evoke a pain response of A-Delta and C fibers. In addition the rate of stimulation can be rapid to lead to the effect of temporal summation. When used with an EEG recording system, a patient's responses to pain perception and evoked potentials (EPs) can be recorded, which provide objective information about integrity of the nociceptive afferents of peripheral nerve system, spinal cord, as well as the brain response of different structures. The CHEPS provide the investigators a practical and convenient tool in clinical application to study pain. The investigators will use the CHEPS as stimulation for studying the heat evoked potentials and analyze the difference between the normal subjects and patients with peripheral nerve diseases. These might help to clarify the mechanism of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with peripheral nerve diseases or other neurological diseased with sensory disturbance
* Normal subjects without:

  * Systemic disease like diabetes mellitus, renal disease or other systemic diseases
  * Abnormal neurological symptoms or signs
  * Psychological disease like affective disorders or psychosis.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Tsang Hsieh, PhD, Study Director — Department of Anatomy and Cell Biology, National Taiwan University College of Medicine; Department of Neurology, National Taiwan University Hospital.
Locations (1):
- Department of Anatomy and Cell Biology, National Taiwan University College of Medicine, Taipei, Taiwan